CLINICAL TRIAL: NCT03522259
Title: BARIVA:Short Versus Extended Prophylaxis of Rivaroxaban for Venous Thromboembolism After Bariatric Surgery
Brief Title: Rivaroxaban as Thrombosis Prophylaxis in Bariatric Surgery
Acronym: BARIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bayer (Industry); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UVCMBS003
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Bariatric Surgery
Keywords: Rivaroxaban; Thromboembolic prophylaxis; Venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Rivaroxaban short arm (Active Comparator): 7 day prophylactic postop treatment after Bariatric surgery with 10mg Rivaroxaban p.o.
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto]
- B: Rivaroxaban long arm (Active Comparator): 28 day prophylactic postop treatment after Bariatric surgery with 10mg Rivaroxaban p.o.
  Subgroup: PK/PD parameters are assessed following the last intake of Rivaroxaban at day 28
  Interventions: Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto]

INTERVENTIONS:
Drug: Rivaroxaban 10 MG Oral Tablet [Xarelto] — Rivaroxaban 10mg per os is started on the first postoperative day. Patients receive Rivaroxaban 10mg QD for 7days (short arm) or 28 days (long arm)

SUMMARY:
The aim of this study is to investigate the efficacy and safety of rivaroxaban in obese patients undergoing bariatric surgery.

The objectives are to assess the safety and feasibility of venous thromboembolism (VTE) prophylaxis and lung embolism with Rivaroxaban 10mg as an oral anticoagulant. After bariatric surgery patients receive the study medication Xarelto 10mg QD for 7, resp. 28 days.

All clinically thromboembolic events will be assessed by ultrasound or CT, respectively, as soon as apparent. In addition, patients are screened for VTE at day 28 by ultrasound to detect clinically inapparent thromboses.

In a subgroup of study patients (patients from the University Hospital Inselspital, Bern) PK/PD parameters are assessed following the last intake of rivaroxaban at day 28.

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy and safety of rivaroxaban in obese patients undergoing bariatric surgery.

Rivaroxaban as an oral anticoagulant could be an attractive option for thromboprophylaxis compared to subcutaneous standard treatment after bariatric surgery. Especially in high-risk patients where an extended duration of thromboprophylaxis after hospital discharge is recommended, an oral therapy would be desirable.

The objectives are to assess the safety and feasibility of VTE prophylaxis and lung embolism with Rivaroxaban 10mg as an oral anticoagulant. Especially in high-risk patients where an extended duration of thromboprophylaxis after hospital discharge is recommended, an oral therapy would be desirable.

After bariatric surgery patients receive the study medication Xarelto 10mg QD for 7, resp. 28 days.

In a subgroup of study patients (patients from the University Hospital Inselspital, Bern) PK/PD parameters are assessed following the last intake of rivaroxaban at day 28.

ELIGIBILITY:
Inclusion Criteria:

* Patients with scheduled elective bariatric surgery or redo surgery after bariatric interventions
* Written informed consent

Exclusion Criteria:

* DVT and/or PE in the patient history
* Myocardial infarction, transient ischemic attack or stroke within 6 months of study entry
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with symptomatic or asymptomatic VTE | 28 days
  Assessed by ultrasound

SECONDARY OUTCOMES:
Number of patients with symptomatic VTE within 28 days after bariatric surgery | 28 days
  Assessed by ultrasound
Number of patients with asymptomatic VTE within 28 days after bariatric surgery | 28 days
  Assessed by ultrasound
All cause mortality within 28 days after bariatric surgery | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Guido Stirnimann, MD, Principal Investigator — Berne, University Hospital, University of Berne, Switzerland
Locations (3):
- Switzerland (3):
  - Kantonsspital Baden, Baden
  - University Hospital, Inselspital Berne, Bern
  - Clinic Beau-Site, Bern

REFERENCES:
- [Derived] Kroll D, Nett PC, Rommers N, Borbely Y, Deichsel F, Nocito A, Zehetner J, Kessler U, Fringeli Y, Alberio L, Candinas D, Stirnimann G. Efficacy and Safety of Rivaroxaban for Postoperative Thromboprophylaxis in Patients After Bariatric Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2315241. doi: 10.1001/jamanetworkopen.2023.15241. PMID 37227726
- [Derived] Amaral FC, Baptista-Silva JC, Nakano LC, Flumignan RL. Pharmacological interventions for preventing venous thromboembolism in people undergoing bariatric surgery. Cochrane Database Syst Rev. 2022 Nov 22;11(11):CD013683. doi: 10.1002/14651858.CD013683.pub2. PMID 36413425